CLINICAL TRIAL: NCT01589900
Title: The Role of Sox2 in Tumor Genesis and Migration in Colorectal Cancer
Brief Title: Identification the Expression of Sox2 in Colorectal Cancer Tissues
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Lixiao Xu, Laboratory of Cancer and Stem Cell Biology, Sun Yat-sen University
Other Study IDs: SYSU
Record Dates: First submitted 2012-04-30; First posted 2012-05-02 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; invasion; metastasis; IHC
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Sox2 has been studied in several types of human solid tumors. The investigators found that Sox2 had higher expression level in colorectal cancer and metastatic tissues than normal tissues. So the investigators assumed that whether Sox2 plays an important role in the progression and migration of colon cancer.

DETAILED DESCRIPTION:
In our study, we examined Sox2 expression in archived human colon cancer tissues and found that its Sox2 expression correlates with reduced patient survival, increased tumor grade and metastasis probability.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of colorectal cancer

Exclusion Criteria:

* Clinical diagnosis characteristics not exactly described in the patients information

Ages: 24 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All rchived 136 tissues were obtained and pathologically confirmed from patients who underwent surgical resections between 2005 and 2006 at the Cancer Center of Sun Yat-sen University (Guangzhou, Guangdong, P. R. China)). The patients from whom the samples were derived underwent curative resection between 2005 and 2006. Tumor differentiation was characterized according to WHO classification, while the surgical pathologic stage was analyzed according to the TNM classification system of the International Union against Cancer. All samples were anonymously coded in accordance with local ethical guidelines.
Sampling Method: Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2005-01; Primary Completion 2006-12 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zhang, M.D.Ph.D, Principal Investigator — Laboratory of Cancer and Stem Cell Biology School of Life Sciences Sun Yat-sen University